CLINICAL TRIAL: NCT00697593
Title: A Phase IV Open Label Study in Moderate to Severe Chronic Plaque Psoriasis Subjects Transitioning From Previous Systemic Antipsoriasis Therapies (Methotrexate, Cyclosporine, Retinoids or Psoralen-Ultraviolet Light A (PUVA), Narrow-Band Ultraviolet Light B (NBUVB) to Raptiva 1mg/kg/ Week Therapy.
Brief Title: ChangE From Any Systemic psoriasiS therapY to Raptiva
Acronym: EASY
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated after the European Medicines Agency recommended to suspend the marketing authorisation of Raptiva in the European Union
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Maria Koutsopoulou, Merck Serono International S.A., an affiliate of Merck KGaA, Darmstadt, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 27809
Record Dates: First submitted 2008-06-11; First posted 2008-06-16 (Estimated); Results first posted 2010-08-30 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Plaque Psoriasis
Keywords: Efalizumab; Chronic Plaque Psoriasis; Transition from systemic therapies on to Efalizumab

ARMS (1):
- Efalizumab (Experimental)
  Interventions: Drug: Efalizumab - anti CD11a recombinant human monoclonal antibody (mAb)

INTERVENTIONS:
Drug: Efalizumab - anti CD11a recombinant human monoclonal antibody (mAb) — Each subject will receive an initial conditioning dose of 0.7 mg/kg/week and then will continue treatment at a dose of 1mg/kg/week for up to 12 weeks.

SUMMARY:
To assess the safety of transitioning subjects to Raptiva therapy from standard oral systemic or phototherapy by overlapping with Raptiva whilst tapering the initial systemic therapy or phototherapy dose.

ELIGIBILITY:
Inclusion Criteria:

1. Are at least 18 years old.
2. Have plaque psoriasis with an sPGA score of at least moderate or severe at time of initiation of previous systemic treatment.
3. Are transitioning from methotrexate, cyclosporine, retinoids, PUVA or NBUVB and initiating treatment with Raptiva according to the decision of the investigator and in accordance with the indication and the recommendations of the Raptiva Investigator Brochure, i.e. to which they have failed to respond, have a contraindication to or are intolerant of other systemic therapies.
4. Agree to participate in the study, and to disclose any medical events to the investigator. The subject must be willing and able to comply with the protocol requirements for the duration of the study.
5. Have given written informed consent with the understanding that consent may be withdrawn at any time without prejudice to future medical care.
6. Women of childbearing potential must use appropriate contraception during treatment and up to the last study visit (safety follow-up visit). For men, it is also mandatory to practice contraception during participation in the trial, as there are no existing data on the effect of Raptiva on spermatogenesis.
7. Discontinuation of any investigational drug or treatment 3 months prior to study start or as per washout requirements from previous protocol.

No primary vaccinations (e.g., tetanus, booster, influenza vaccine) for at least 14 days prior to first dose of study drug.For the purposes of this trial, women of childbearing potential is defined as: "All female subjects after puberty unless they are post-menopausal for at least two years, are surgically sterile or are sexually inactive."

Exclusion Criteria:

1. Any contra-indication to Raptiva, according to the Investigator Brochure, or as follows:

   * Hypersensitivity to Raptiva or to any of the excipients.
   * Subjects with history of malignancies.
   * History of active tuberculosis (TB) or currently undergoing treatment for TB. Purified Protein Derivative (PPD) testing or chest X-ray is required for high-risk subjects. Subjects with a positive PPD (not due to BCG vaccination) or chest X-ray will be excluded.
   * Subjects with specific forms of psoriasis like guttate, erythrodermic or pustular psoriasis as sole or predominant form of psoriasis.
   * Subjects with immunodeficiencies.
2. Simultaneous participation in another clinical trial.
3. Subjects experiencing a psoriasis exacerbation during screening period.
4. Subjects who have previously been on Raptiva treatment who withdrew due to lack of efficacy or an adverse event. If withdrawal was due to another non-drug reason (vaccination, or infection) then the subject can be included in this study.
5. History of hepatitis B, hepatitis C or human immunodeficiency virus (HIV).
6. History of thrombocytopenia, haemolytic anaemia or clinically significant anaemia.
7. Hepatic enzyme levels =/>3 times the upper limit of normal or serum creatinine level =/>2 times the upper limit of normal.
8. Pregnant or breast-feeding.
9. Any medical condition (prior or existing) that, in the judgment of the investigator or sponsor, could jeopardize the subject's safety following exposure to study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Selenko-Gebauer, Study Director — Merck Serono International S.A., an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Probity Medical Research, City Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of first subject first visit: 22 January 2008 Date of last subject last visit: 21 April 2009 Subjects were enrolled at 13 study centers in 2 countries, including 10 study centers in Canada and 3 study centers in the Netherlands.
Pre-assignment Details: Subjects were to be screened for study eligibility within 14 days before Day 1
Groups:
- Efalizumab: Each subject received an initial conditioning dose of efalizumab of 0.7 mg/kg/week and then was to continue treatment at a dose of 1 mg/kg/week for up to 12 weeks. Efalizumab was administered by subcutaneous injection
Period: Overall Study
Arm/Group | Efalizumab
Started | 70
Completed | 51
Not Completed | 19
Not completed — Adverse Event | 3
Not completed — Protocol Violation | 1
Not completed — Lack of Efficacy | 3
Not completed — Suspension of the study by sponsor | 12

BASELINE CHARACTERISTICS:
Arm/Group | Efalizumab
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (14.7)
Age, Customized [Number; unit: participants]
  18 - 40 years | 26
  41 to 64 years | 36
  >64 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 45
Region of Enrollment [Number; unit: participants]
  Canada | 60
  Netherlands | 10
static Physician's Global Assessment (sPGA) [Number; unit: participants] — Numbers of participants with sPGA ratings of clear; minimal; mild; moderate; severe; or very severe
  participants
    Clear | 0
    Minimal | 4
    Mild | 6
    Moderate | 38
    Severe | 21
    Very Severe | 1
Biochemistry - C-Reactive Protein (CRP) [Number; unit: participants] — Numbers of participants with CRP values <3 mg/L, 3-6 mg/L, and >6 mg/L
  participants
    Participants with <3 mg/L | 36
    Participants with 3 mg/L-6mg/L | 19
    Participants with >6 mg/L | 15
Biochemistry - Alanine Transaminase (ALT) [Mean (Standard Deviation); unit: IU/L] | 27.8 (12.2)
Biochemistry - Alkaline Phosphatase [Mean (Standard Deviation); unit: IU/L] | 76.6 (19.0)
Biochemistry - Aspartate Transaminase (AST) [Mean (Standard Deviation); unit: IU/L] | 23.0 (7.8)
Biochemistry - Creatinine [Mean (Standard Deviation); unit: μmol/L] | 82.9 (18.9)
Biochemistry - Glutamyl Transferase [Mean (Standard Deviation); unit: IU/L] | 25.9 (15.3)
Biochemistry - Potassium [Mean (Standard Deviation); unit: mmol/L] | 4.19 (0.36)
Biochemistry - Values: Sodium [Mean (Standard Deviation); unit: mmol/L] | 139.5 (1.9)
Biochemistry - Total Bilirubin [Mean (Standard Deviation); unit: μmol/L] | 8.0 (4.7)
Biochemistry - Urea [Mean (Standard Deviation); unit: mmol/L] | 5.677 (1.633)
Hematology - Hematocrit [Mean (Standard Deviation); unit: packed cell volume] | 0.430 (0.040)
Hematology - Hemoglobin [Mean (Standard Deviation); unit: g/L] | 145.0 (13.7)
Hematology - Red Blood Cell Count [Mean (Standard Deviation); unit: x10^12/L] | 4.69 (0.52)
Hematology - White Blood Cell Count [Mean (Standard Deviation); unit: x10^9/L] | 7.11 (1.95)
Hematology - Basophils [Mean (Standard Deviation); unit: x10^9/L] | 0.032 (0.033)
Hematology - Eosinophils [Mean (Standard Deviation); unit: x10^9/L] | 0.177 (0.135)
Hematology - Lymphocytes [Mean (Standard Deviation); unit: x10^9/L] | 1.911 (0.670)
Hematology - Monocytes [Mean (Standard Deviation); unit: x10^9/L] | 0.462 (0.188)
Hematology - Neutrophils [Mean (Standard Deviation); unit: x10^9/L] | 4.533 (1.582)
Hematology - Platelet Count [Mean (Standard Deviation); unit: x10^9/L] | 256.0 (54.7)
Urinalysis - Glucose [Number; unit: participants] — Number of participants with or without glucose detected in urine
  participants
    Negative | 66
    Present | 4
Urinalysis - Ketones [Number; unit: participants] — Number of participants with or without ketones detected in urine
  participants
    Negative | 67
    Present | 3
Urinalysis - Values - Nitrite [Number; unit: participants] — Number of participants with or without nitrite detected in urine
  participants
    Negative | 69
    Positive | 1
Urinalysis - Leukocytes Esterase [Number; unit: participants] — Number of participants with or without leukocytes esterase detected in urine
  participants
    Negative | 60
    Present | 10
Urinalysis - Values - Protein [Number; unit: participants]
  Negative | 59
  Present | 11
Urinalysis - Blood [Number; unit: participants] — Number of participants with or without blood detected in urine
  participants
    Negative | 66
    Present | 4
Urinalysis - pH [Mean (Standard Deviation); unit: pH units] | 5.84 (0.49)

OUTCOME MEASURES:

1. Primary Outcome: Hematology - Hematocrit
Description: Blood samples were taken for clinical laboratory testing
Time Frame: Week 12 / Early Termination
Population: Safety Population - 4 participants missing values
Measure: Mean (Standard Deviation); unit: packed cell volume
Arm/Group | Efalizumab
Number analyzed (Participants) | 66
packed cell volume | 0.434 (0.039)

2. Secondary Outcome: Static Physician's Global Assessment (sPGA)
Description: Number of subjects who achieve an Static Physician's Global Assessment (sPGA) rating of clear; minimal; mild; moderate; severe; or very severe at Week 12 (Day 85).
Time Frame: 12 Weeks/Early Termination
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Efalizumab
Number analyzed (Participants) | 69
participants
  Clear | 3
  Minimal | 19
  Mild | 20
  Moderate | 21
  Severe | 6
  Very Severe | 0

3. Primary Outcome: Hematology - Hemoglobin
Description: Blood samples were taken for clinical laboratory testing
Time Frame: Week 12 / Early Termination
Population: Safety Population - 3 participants missing values
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Efalizumab
Number analyzed (Participants) | 67
g/L | 144.8 (13.0)

4. Primary Outcome: Hematology - Red Blood Cell Count
Description: Blood samples were taken for clinical laboratory testing
Time Frame: Week 12 / Early Termination
Population: Safety Population - 3 participants missing values
Measure: Mean (Standard Deviation); unit: x10^12/L
Arm/Group | Efalizumab
Number analyzed (Participants) | 67
x10^12/L | 4.78 (0.52)

5. Primary Outcome: Hematology - White Blood Cell Count
Description: Blood samples were taken for clinical laboratory testing
Time Frame: Week 12 / Early Termination
Population: Safety Population - 3 participants missing values
Measure: Mean (Standard Deviation); unit: x10^9/L
Arm/Group | Efalizumab
Number analyzed (Participants) | 67
x10^9/L | 10.06 (2.69)

6. Primary Outcome: Hematology - Neutrophils
Description: Blood samples were taken for clinical laboratory testing
Time Frame: Week 12 / Early Termination
Population: Safety Population - 3 participants missing values
Measure: Mean (Standard Deviation); unit: x10^9/L
Arm/Group | Efalizumab
Number analyzed (Participants) | 67
x10^9/L | 5.047 (1.976)

7. Primary Outcome: Hematology - Eosinophils
Description: Blood samples were taken for clinical laboratory testing
Time Frame: Week 12 / Early Termination
Population: Safety Population - 3 participants missing values
Measure: Mean (Standard Deviation); unit: x10^9/L
Arm/Group | Efalizumab
Number analyzed (Participants) | 67
x10^9/L | 0.206 (0.130)

8. Primary Outcome: Hematology - Basophils
Description: Blood samples were taken for clinical laboratory testing
Time Frame: Week 12 / Early Termination
Population: Safety Population - 3 participants missing values
Measure: Mean (Standard Deviation); unit: x10^9/L
Arm/Group | Efalizumab
Number analyzed (Participants) | 67
x10^9/L | 0.050 (0.038)

9. Primary Outcome: Hematology - Monocytes
Description: Blood samples were taken for clinical laboratory testing
Time Frame: Week 12 / Early Termination
Population: Safety Population - 3 participants missing values
Measure: Mean (Standard Deviation); unit: x10^9/L
Arm/Group | Efalizumab
Number analyzed (Participants) | 67
x10^9/L | 0.526 (0.205)

10. Primary Outcome: Hematology - Lymphocytes
Description: Blood samples were taken for clinical laboratory testing
Time Frame: Week 12 / Early Termination
Population: Safety Population - 3 participants missing values
Measure: Mean (Standard Deviation); unit: x10^9/L
Arm/Group | Efalizumab
Number analyzed (Participants) | 67
x10^9/L | 4.209 (1.220)

11. Primary Outcome: Hematology - Platelet Count
Description: Blood samples were taken for clinical laboratory testing
Time Frame: Week 12 / Early Termination
Population: Safety Population - 4 participants missing values
Measure: Mean (Standard Deviation); unit: x10^9/L
Arm/Group | Efalizumab
Number analyzed (Participants) | 66
x10^9/L | 255.5 (64.8)

12. Primary Outcome: Biochemistry - Sodium
Description: Blood samples were taken for clinical laboratory testing
Time Frame: Week 12 / Early Termination
Population: Safety Population - 1 participant missing values
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Efalizumab
Number analyzed (Participants) | 69
mmol/L | 139.0 (2.1)

13. Primary Outcome: Biochemistry - Potassium
Description: Blood samples were taken for clinical laboratory testing
Time Frame: Week 12 / Early Termination
Population: Safety Population - 1 participant missing values
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Efalizumab
Number analyzed (Participants) | 69
mmol/L | 4.23 (0.41)

14. Primary Outcome: Biochemistry - Creatinine
Description: Blood samples were taken for clinical laboratory testing
Time Frame: Week 12 / Early Termination
Population: Safety Population - 1 participant missing values
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Efalizumab
Number analyzed (Participants) | 69
μmol/L | 83.1 (20.1)

15. Primary Outcome: Biochemistry - Total Bilirubin
Description: Blood samples were taken for clinical laboratory testing
Time Frame: Week 12 / Early Termination
Population: Safety Population - 1 participant missing values
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Efalizumab
Number analyzed (Participants) | 69
μmol/L | 7.2 (3.7)

16. Primary Outcome: Biochemistry - Aspartate Transaminase (AST)
Description: Blood samples were taken for clinical laboratory testing
Time Frame: Week 12 / Early Termination
Population: Safety Population - 2 participants missing values
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Efalizumab
Number analyzed (Participants) | 68
IU/L | 22.2 (9.6)

17. Primary Outcome: Biochemistry - Alanine Transaminase (ALT)
Description: Blood samples were taken for clinical laboratory testing
Time Frame: Week 12 / Early Termination
Population: Safety Population - 1 participant missing values
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Efalizumab
Number analyzed (Participants) | 69
IU/L | 28.7 (19.3)

18. Primary Outcome: Biochemistry - Alkaline Phosphatase
Description: Blood samples were taken for clinical laboratory testing
Time Frame: Week 12 / Early Termination
Population: Safety Population - 1 participant missing values
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Efalizumab
Number analyzed (Participants) | 69
IU/L | 80.2 (21.1)

19. Primary Outcome: Biochemistry - Glutamyl Transferase
Description: Blood samples were taken for clinical laboratory testing
Time Frame: Week 12 / Early Termination
Population: Safety Population - 1 participant missing values
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Efalizumab
Number analyzed (Participants) | 69
IU/L | 28.6 (20.1)

20. Primary Outcome: Biochemistry - Urea
Description: Blood samples were taken for clinical laboratory testing
Time Frame: Week 12 / Early Termination
Population: Safety Population - 1 participant missing values
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Efalizumab
Number analyzed (Participants) | 69
mmol/L | 5.283 (1.628)

21. Primary Outcome: Biochemistry - C-Reactive Protein (CRP)
Description: Blood samples were taken for clinical laboratory testing of the numbers of participants with CRP values <3 mg/L, 3-6 mg/L, and >6 mg/L
Time Frame: Week 12 / Early Termination
Population: Safety Population - 1 participant with missing values
Measure: Number; unit: participants
Arm/Group | Efalizumab
Number analyzed (Participants) | 69
participants
  participants with <3 mg/L | 28
  participants with 3-6 mg/L | 22
  participants with >6 mg/L | 19

22. Primary Outcome: Urinalysis - pH
Description: Urine samples were taken for clinical laboratory testing
Time Frame: Week 12 / Early Termination
Population: Safety Population - 3 participants missing values
Measure: Mean (Standard Deviation); unit: pH units
Arm/Group | Efalizumab
Number analyzed (Participants) | 67
pH units | 5.75 (0.47)

23. Primary Outcome: Urinalysis - Protein
Description: Urine samples were taken for clinical laboratory testing of the number of participants with or without protein in urine
Time Frame: Week 12 / Early Termination
Measure: Number; unit: participants
Arm/Group | Efalizumab
Number analyzed (Participants) | 67
participants
  Negative | 54
  Present | 13

24. Primary Outcome: Urinalysis - Ketones
Description: Urine samples were taken for clinical laboratory testing of the number of participants with or without ketones in urine
Time Frame: Week 12 / Early Termination
Measure: Number; unit: participants
Arm/Group | Efalizumab
Number analyzed (Participants) | 67
participants
  Negative | 58
  Present | 9

25. Primary Outcome: Urinalysis - Glucose
Description: Urine samples were taken for clinical laboratory testing of the number of participants with or without glucose in urine
Time Frame: Week 12 / Early Termination
Population: Safety Population - 3 participants with missing values
Measure: Number; unit: participants
Arm/Group | Efalizumab
Number analyzed (Participants) | 67
participants
  Negative | 64
  Present | 3

26. Primary Outcome: Urinalysis - Blood
Description: Urine samples were taken for clinical laboratory testing of the number of participants with or without blood in urine
Time Frame: Week 12 / Early Termination
Population: Safety Population - 3 participants with missing values
Measure: Number; unit: participants
Arm/Group | Efalizumab
Number analyzed (Participants) | 67
participants
  Negative | 58
  Present | 9

27. Primary Outcome: Urinalysis - Nitrite
Description: Urine samples were taken for clinical laboratory testing of the number of participants with or without nitrite in urine
Time Frame: Week 12 / Early Termination
Population: Safety Population - 3 participants with missing values
Measure: Number; unit: participants
Arm/Group | Efalizumab
Number analyzed (Participants) | 67
participants
  Negative | 65
  Positive | 2

28. Primary Outcome: Urinalysis - Leukocytes Esterase
Description: Urine samples were taken for clinical laboratory testing of the number of participants with or without leukocytes esterase in urine
Time Frame: Week 12 / Early Termination
Population: Safety Population - 3 participants with missing values
Measure: Number; unit: participants
Arm/Group | Efalizumab
Number analyzed (Participants) | 67
participants
  Negative | 60
  Present | 7

29. Primary Outcome: Adverse Events, Serious Adverse Events, and Laboratory Data (Haematology and Biochemistry) and Urinalysis
Description: Information on adverse events are displayed in the adverse events section. Information laboratory data and urinalysis findings are displayed individually above
Time Frame: Week 12 / Early Termination
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 Weeks
Description: 'Other Adverse Events' table shows the number of participants experiencing any adverse event and the listing shows all treatment emergent adverse events occuring above the threshold value in the Safety Population
Arm/Group | Efalizumab
Serious Adverse Events (participants affected / at risk) | 0/70
Other Adverse Events (participants affected / at risk) | 50/70
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Efalizumab (N=70)
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Candidiasis (Infections and infestations) | 1
Chills (General disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dermal cyst (Skin and subcutaneous tissue disorders) | 3
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 3
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Epilepsy (Nervous system disorders) | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 3
Flushing (Vascular disorders) | 1
Folliculitis (Infections and infestations) | 2
Furuncle (Infections and infestations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Gastroenteritis (Infections and infestations) | 1
Gout (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 10
Heart rate increased (Investigations) | 1
Hot flush (Vascular disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Influenza (Infections and infestations) | 4
Influenza like illness (General disorders) | 5
Lower respiratory tract infection (Infections and infestations) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nasopharyngitis (Infections and infestations) | 5
Nausea (Gastrointestinal disorders) | 1
Oral herpes (Infections and infestations) | 1
Orthostatic hypotension (Vascular disorders) | 1
Otitis media (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 4
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1
Sciatica (Nervous system disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Sinusitis (Infections and infestations) | 1
Sweat gland infection (Infections and infestations) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 2
Upper respiratory tract infection (Infections and infestations) | 8
Urinary tract infection (Infections and infestations) | 2
Vascular occlusion (Vascular disorders) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Conjunctivitis (Eye disorders) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other